CLINICAL TRIAL: NCT05850455
Title: A Comparative Study Between Lumbar Epidural Analgesia Versus Local Analgesia With Dexmedetomidine Infusion in Endoscopic Lumbar Discectomy
Brief Title: Lumbar Epidural Analgesia Versus Local Anesthesia With Dexmedetomidine Infusion in Endoscopic Lumbar Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAMSU R 280/2022/2023
Record Dates: First submitted 2023-04-19; First posted 2023-05-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Bupivacaine; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): will receive local anesthesia with dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine Hydrochloride 'Precedex' combined with; Drug: Local infiltration with Lidocaine HCL 1%'Debocaine'
- Group B (Experimental): will receive epidural analgesia
  Interventions: Procedure: Lumbar epidural analgesia with Bupivacaine 0.25% 'Sunnypivacaine'
- Group Con (Experimental): will receive general anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride 'Precedex' combined with — Dexmedetomidine Hydrochloride which is an Alfa 2 receptor agonist
  Arms: Group A
Procedure: Lumbar epidural analgesia with Bupivacaine 0.25% 'Sunnypivacaine' — The epidural insertion point will be 2 segments upper than the surgical procedure level, 10 ml of Bupivacaine 0.25% will be injected in the epidural space to adjust the sensory level
  Arms: Group B
Procedure: General anesthesia — Propofol 2-3 mg/kg'Diprivan 1%', Fentanyl 'Fentanyl' 2 μg/kg, and Cisatracurium 'Cisatracure' 0.2 mg/kg will be administered to facilitate endotracheal intubation, and ventilation will be controlled to maintain the end-tidal carbon dioxide (CO2) between 32-38 mmHg, to maintain anesthesia, 2-3% Sevoflurane 'Sevoflurane', and 0.05 mg/kg of the muscle relaxant Cisatracurium will be added at 40-minute intervals according to the conditions of the operation. No other medication will be administered
  Arms: Group Con
Drug: Local infiltration with Lidocaine HCL 1%'Debocaine' — Lidocaine 1% which is a local analgesic as local infiltration
  Arms: Group A

SUMMARY:
To compare between local anesthesia combined with intravenous Dexmedetomidine and epidural analgesia as regard the effectiveness and patient satisfaction during percutaneous transforaminal endoscopic discectomy.

DETAILED DESCRIPTION:
Percutaneous transforaminal endoscopic discectomy. under LA is recommended in consideration of safety. Under LA, patients keep conscious during the process of PTED, and the surgeon can obtain feedback directly from the patients if the nerve is interfered. Dexmedetomidine, a highly selective alpha 2 adrenoreceptor agonist, has unique characteristics in providing sedation and analgesia. Due to its central sympatholytic action, Dexmedetomidine produces dose-dependent sedation, antinociception and anxiolysis. Epidural anesthesia is another major method which can keep patients awake during surgery and the surgeons can check the function of the nerve from the maintained motor function of patients' lower limbs

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to II.
2. Aged 18 to 50 years.
3. Both sexes.

Exclusion Criteria:

* Spinal malformation
* Recurrent LDH
* Multi segment LDH
* Patients younger than 18 years or older than 50 years
* Patients with hypersensitivity to one of the used drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS), A score from 0 -10 where 10indicates the worst pain possible | 4 hours
  The first outcome is to compare the VAS preoperative, intraoperative for group A, B and 1 hour postoperative for group A, B and Con
Heart rate | 9 hours
  Comparing the Heart rate ( Heart beats per minute) for the 3 groups every 30 minutes intraoperative and every hour postoperative for 6 hours
Postoperative anesthetic complications | 2 days
  Assess and compare postoperative anesthetic complications postoperative, 1 day postoperative and 2 days postoperative
Satisfaction rate of anesthesia | 1 hour
  To compare satisfaction rate of anesthesia 1 hour postoperative Using the .The Heidelberg Peri-anaesthetic Questionnaire
Systolic and Diastolic Blood pressure | 9 hours
  Comparing the systolic and diastolic Blood Pressure in mmHG for the 3 groups every 30 minutes intraoperative and every hour postoperative for 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No